CLINICAL TRIAL: NCT06555354
Title: MicroRNAs Methylation and Expression Profiling for Identification of Breast Cancer Patients at High Risk to Develop Distant Metastases
Brief Title: MicroRNAs and Prognosis in Breast Cancer
Acronym: BREMIR
Status: Completed | Type: Observational
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Principal Investigator, Paola Parrella, Medical Doctor, Casa Sollievo della Sofferenza IRCCS
Other Study IDs: BREMIR
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female; Metastases Breast
Keywords: microRNA; prognosis; risk prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — RNA and DNA obtained from fresh frozen and/or FFPE tissues Plasma Sample for miRNA analyses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Identification in a retrospective cohort of a miRNA panel associated with the development of distant metastases.The retrospective cohort consists of tumor and normal tissue obtained from breast cancer patients, stored at -80°C at the Laboratory of Oncology. Of these samples, 360 met the inclusion criteria.
  Interventions: Diagnostic Test: miRNA targeted analysis on breast cancer tissues; Diagnostic Test: miRNA profiling of breast cancer tissues
- Prospective: The association between miRNA expression and the clinical course of the disease identified in the retrospective cohort, is being confirmed in an independent prospective cohort. Both normal and tumor tissues of the patients, as well as plasma collected before surgery and at each follow-up time point, is being analyzed. Based on the annual number of surgeries performed at the Breast Surgery Unit, we initially estimated that the prospective cohort would consist of about 500 patients recruited over three years. Since the project was extended for additional two years the actual number of subject recruited was 972. In addition plasma sample for 100 breast benign condition was also collected as controls.
  Interventions: Diagnostic Test: miRNA targeted analysis on breast cancer tissues; Diagnostic Test: miRNA targeted analysis on plasma samples

INTERVENTIONS:
Diagnostic Test: miRNA targeted analysis on breast cancer tissues — Total RNA is extracted from tissue sample and selected miRNA quantified by PCR based relative quantification method (QPCR) with a standard curve.
Diagnostic Test: miRNA targeted analysis on plasma samples — miRNAs extracted from plasma samples are analysed by QPCR and/or ddPCR .
  Groups: Prospective
Diagnostic Test: miRNA profiling of breast cancer tissues — Selected samples from the retrospective cohort are profiled for miRNA expression by using GeneChip® miRNA 4.0 Array.
  Groups: Retrospective

SUMMARY:
Mono-centric, observational retrospective and prospective study, designed for breast cancer patients to identify novel miRNA based biomarker able to predict metastases development in breast cancer patients.

DETAILED DESCRIPTION:
The potential role of miRNAs will be studied as a predictor of metastases development. miRNAs expression and miRNAs promoter methylation will be evaluated in surgically removed specimens obtained from breast cancer patients at diagnosis. Relevant miRNAs will be first identified by analysing a retrospective breast cancer cohort including at least and subsequently validated on a prospective cohort.

ELIGIBILITY:
Retrospective Cohort

Inclusion Criteria:

Tissue samples from breast cancer cases diagnosed from 2004 to 2014 for which informed consent for tumour banking and complete clinicopathological and follow up data were available.

Exclusion Criteria:

Pre-surgery neoadjuvant treatment for breast cancer with chemotherapy, lapatinib, trastuzumab, letrozole, anastrozole, exemestane or tamoxifen.

Other cancers diagnosed in the last five years.

Prospective Cohort:

Inclusion Criteria:

Ability to provide written informed consent; Age greater than 18 years; Histological diagnosis of Breast disease; First diagnosis of Breast Cancer; Syncronous distant metastasis absent.

Exclusion Criteria:

Stage IV breast cancer; Pre-surgery neoadjuvant treatment for breast cancer with chemotherapy, lapatinib, trastuzumab, letrozole, anastrozole, exemestane or tamoxifen; Other cancers diagnosed in the last five years; Alteration of mental status, dementia, or any psychiatric condition that might impair the ability to consciously sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective Cohort: 260 patients diagnosed with breast cancer of any histological type that underwent surgery for breast cancer from 2004 to 2014. For all this subjects fresh frozen specimen collected at the time of surgery are available for DNA and/or RNA extraction.
  Prospective cohort: 1072 individuals were enrolled in this study from December 2014 to December 2019: 972 patients were affected by breast cancer, 100 patients showed benign breast lesions. For all this subjects fresh frozen specimen and/or FFPE sample at diagnosis, together with a plasma sample collected at the time of surgery are available for DNA and/or RNA extraction. For invasive breast cancer at least two plasma samples were colleted at surgery and after surgery. A third plasma sample is being collected at the eventual progression.
Sampling Method: Non-Probability Sample
Enrollment: 1432 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Risk of metastases development | evaluation 5 and 10 years after diagnosis
  Identification of miRNAs associated with the risk to develop distant metastases.

SECONDARY OUTCOMES:
Overall Survival | evaluation 5 and 10 years after diagnosis
  Identification of miRNAs associated with the risk of cancer specific death

CONTACTS AND LOCATIONS:
Locations (1):
- Casa sollievo della Sofferenza IRCCS, San Giovanni Rotondo, FG, Italy

REFERENCES:
- [Background] Barbano R, Pasculli B, Rendina M, Fontana A, Fusilli C, Copetti M, Castellana S, Valori VM, Morritti M, Graziano P, Luigi C, Coco M, Picardo F, Mazza T, Evron E, Murgo R, Maiello E, Esteller M, Fazio VM, Parrella P. Stepwise analysis of MIR9 loci identifies miR-9-5p to be involved in Oestrogen regulated pathways in breast cancer patients. Sci Rep. 2017 Mar 27;7:45283. doi: 10.1038/srep45283. PMID 28345661
- [Background] Pasculli B, Barbano R, Fontana A, Biagini T, Di Viesti MP, Rendina M, Valori VM, Morritti M, Bravaccini S, Ravaioli S, Maiello E, Graziano P, Murgo R, Copetti M, Mazza T, Fazio VM, Esteller M, Parrella P. Hsa-miR-155-5p Up-Regulation in Breast Cancer and Its Relevance for Treatment With Poly[ADP-Ribose] Polymerase 1 (PARP-1) Inhibitors. Front Oncol. 2020 Aug 12;10:1415. doi: 10.3389/fonc.2020.01415. eCollection 2020. PMID 32903519
- [Background] Pasculli B, Barbano R, Rendina M, Fontana A, Copetti M, Mazza T, Valori VM, Morritti M, Maiello E, Graziano P, Murgo R, Fazio VM, Esteller M, Parrella P. Hsa-miR-210-3p expression in breast cancer and its putative association with worse outcome in patients treated with Docetaxel. Sci Rep. 2019 Oct 17;9(1):14913. doi: 10.1038/s41598-019-51581-3. PMID 31624308
- [Background] Fontana A, Barbano R, Dama E, Pasculli B, Rendina M, Morritti MG, Melocchi V, Castelvetere M, Valori VM, Ravaioli S, Bravaccini S, Ciuffreda L, Graziano P, Maiello E, Copetti M, Fazio VM, Esteller M, Bianchi F, Parrella P. Combined analysis of miR-200 family and its significance for breast cancer. Sci Rep. 2021 Feb 3;11(1):2980. doi: 10.1038/s41598-021-82286-1. PMID 33536459
- [Derived] Fontana A, Barbano R, Pasculli B, Mazza T, Palumbo O, Binda E, Trivieri N, Mencarelli G, Laurenzana I, Lamorte D, De Luca L, Caivano A, Biagini T, Rendina M, Lo Mele A, Prencipe G, Bravaccini S, Murgo R, Ciuffreda L, Morritti M, Valori VM, Di Lisa FS, Vici P, Castelvetere M, Carella M, Graziano P, Maiello E, Copetti M, Esteller M, Parrella P. Development of a microRNA-based prognostic model for accurate prediction of distant metastasis in breast cancer patients. Breast Cancer Res. 2025 Sep 29;27(1):170. doi: 10.1186/s13058-025-02124-4. PMID 41024243

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT06555354/Prot_SAP_000.pdf